CLINICAL TRIAL: NCT04725214
Title: Anlotinib Combined With STUPP Protocol as First-line Regimen for MGMT Nonmethylated Glioblastoma: a Multicenter, Open-label, Single-arm, Phase II Clinical Trial
Brief Title: Anlotinib Combined With STUPP for MGMT Nonmethylated Glioblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-780
Record Dates: First submitted 2021-01-17; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: MGMT-Unmethylated Glioblastoma
MeSH Terms: interventions — anlotinib; Temozolomide

STUDY DESIGN:
Intervention Model Description: Adjuvant therapy with Anlotinib and Temozolomide for MGMT nonmethylated glioblastoma after concurrent chemo-radiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): For MGMT unmethylated glioblastoma, during temozolomide adjuvant, concurrent with anti-angiogenesis targeted therapy(Anlotinib capsule,d1-14)
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib With STUPP Regimen
  Other Names: temozolomide capsule

SUMMARY:
The purpose of this study is to test the efficacy and safety of Anlotinib in combination with STUPP regimen for MGMT promoter nonmethylated glioblastoma.

DETAILED DESCRIPTION:
For MGMT unmethylated glioblastoma patients undergoing STUPP regimen adjuvant therapy, during adjuvant chemotherapy, concurrent with anti-angiogenesis targeted therapy(Anlotinib capsule,d1-14).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years,
2. Histologically proven diagnosis of glioblastoma (WHO grade IV),
3. Have received standard STUPP treatment plan,
4. Gross resection or partial resection of the tumor (confirmed by MRI)> 50%,
5. The pathological tissue specimens are detected as MGMT unmethylated,6.Karnofsky performance status ≥ 60,
6. No previous radiotherapy, chemotherapy, immunotherapy or biotherapy 7.Adequate bone marrow function: Hemoglobin ≥ 100g/L，Platelets ≥ 80×109/L，Absolute neutrophil count (ANC) ≥ 1.5×109/L

8.Adequate renal function: Serum creatinine ≤ 1.25 x UNL (upper normal limit) or creatinine clearance ≥ 60 ml/min 9.Adequate hepatic function: serum bilirubin ≤ 1.5 x UNL, AST and ALT ≤ 2.5 x UNL，ALP≤5x UNL 10.For females of child-bearing potential, negative serum pregnancy test within 14 days prior to registration. Women of childbearing potential and male participants must practice adequate contraception during participation in the study and within 8 weeks after the last administration of the drug 11.Able to provide written informed consent

Exclusion Criteria:

1. Recurrent or multiple malignant gliomas
2. Subtentorial glioblastoma or metastatic lesions outside the skull
3. Have received radiotherapy, chemotherapy or other anti-tumor drugs for the disease before surgery
4. Previously received radiation therapy for the head and neck cancer
5. Have received any antibody treatment before
6. Contraindication of radiotherapy and chemotherapy defined as follows: Acute bacterial or fungal infection，Unstable angina and/or congestive heart failure within the last 6 months，co-morbidity with immunosuppressive therapy
7. Evidence of bleeding diathesis or coagulopathy
8. Prior invasive malignancy (except for non-melanomatous skin cancer or carcinoma in situ of cervix)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
1-year OS | from enrollment to death (for any reason).assessed up to 12 months
  1-year overall survival

SECONDARY OUTCOMES:
PFS | from enrollment to progression or death (for any reason),assessed up to 24months
  Progression-Free Survival
OS | from enrollment to death (for any reason).assessed up to 24 months
  Overall Survival
adverse event | from enrollment to death (for any reason).assessed up to 24 months
  Adverse events are described in terms of CTC AE 5.0
Health-related quality of life | from enrollment to death (for any reason).assessed up to 24 months
  Health-related quality of life are measured by the EORTC-QL30/BN20
Neurocognitive function | from enrollment to death (for any reason).assessed up to 24 months
  Neurocognitive function are measured by John-Hopkins adapted cognitive exam (ACE)

CONTACTS AND LOCATIONS:
Overall Officials: Qichun Wei, MD, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No